CLINICAL TRIAL: NCT01877811
Title: An Open-Label, Phase 1/1b, Single-Agent Study of RXDX-105 in Patients With Advanced Solid Tumors
Brief Title: Study of RXDX-105, Potent RET Inhibitor in Patients With Advanced Lung Cancer and Other Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RXDX-105-01
Record Dates: First submitted 2013-05-06; First posted 2013-06-14 (Estimated); Last update posted 2019-04-25 (Actual); Status verified 2019-04

CONDITIONS: Solid Tumors
Keywords: Lung Cancer; RET Inhibitor; Solid Tumors; RET mutations or rearrangements; BRAF mutations or rearrangements; Squamous NSCLC; KRAS mutation; Other Lung adenocarcinomas
MeSH Terms: conditions — Lung Neoplasms | interventions — agerafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- RXDX-105 (Experimental)
  Interventions: Drug: RXDX-105

INTERVENTIONS:
Drug: RXDX-105 — During Phase 1/1b, subjects will receive daily oral doses of RXDX-105 in 28-day cycles (except for Day 2 of Cycle 1). To determine the recommended Phase 2 dose (RP2D), doses will be administered in an escalated fashion starting at 20 mg/day.
  During Phase 1b, subjects will be administered the RP2D in 28-day treatment cycles until documented radiographic progression, unacceptable toxicity, withdrawal of consent, or protocol specified parameters to stop treatment.
  Other Names: CEP-32496, AC013773

SUMMARY:
This is a first-in-human, multicenter, open-label study consisting of 2 phases. Phase 1 is a dose escalation study of RXDX-105 (formerly known as CEP-32496) in patients with advanced solid tumors aimed at defining the recommended Phase 2 dose (RP2D) and schedule for administration. Phase 1b is a dose expansion in approximately 90 patients with advanced solid tumors with specific histologies and/or molecular alterations of interest. Patients in Phase 1b will be treated at the RP2D determined in Phase 1.

DETAILED DESCRIPTION:
The primary objective of Phase 1 is to determine the recommended Phase 2 dose (RP2D) of RXDX-105. The primary objective of Phase 1b is to further assess the safety profile and tolerability of RXDX-105 at the RP2D The secondary objective is to evaluate the antitumor activity of RXDX-105 at the RP2D, as assessed by objective response rate (ORR) (complete response [CR] or partial response [PR]) using Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST v1.1) in patients with advanced solid tumors with RET or BRAF mutations or rearrangements.

The RP2D has been determined and Phase 1 portion of the study is now closed to new patient enrollment.

Phase 1 b is open and enrolling patients with solid tumors harboring a RET rearrangement or mutation, or a BRAF rearrangement or mutation. Additionally, patients with Squamous NSCLC and lung adenocarcinomas with other alterations than RET or BRAF such as KRAS mutations, etc. will also be enrolled. Approximately 90 patients will be enrolled in Phase 1b.

Each phase of this study will consist of a 28-day screening period. Patients will be treated in 28-day treatment cycles until documented radiographic progression, unacceptable toxicity, withdrawal of consent, or protocol specified parameters to stop treatment. Patients in Phase 1 and 1b will be followed for 6 months after the last dose of study treatment.

ELIGIBILITY:
Inclusion Criteria for Phase 1b:

1. Patients must have histologically or cytologically confirmed advanced solid tumors with a histology and/or molecular alteration of interest as defined in Section 4, detected by a CLIA-certified or equivalently accredited diagnostic laboratory

   • Squamous NSCLC and Non-squamous NSCLC (no known RET alterations or BRAF V600E mutations) patients must have archival tissue available for analysis by Ignyta; all other patients must send tissue to Ignyta, if tissue is available
2. Prior Treatment:

   * Patients with BRAF V600E mutations must be TKI-naïve; any number of other prior therapies are allowed
   * NSCLC patients with RET alterations who have had a prior RET inhibitor or are RET inhibitor-naïve will be enrolled; (any number of other prior therapies are allowed); all other histologies with RET alterations must be RET inhibitor-naïve
   * Patients with Squamous NSCLC and Non-squamous NSCLC (no known RET alterations or BRAF V600E mutations) may have had prior TKIs and any number of other prior therapies
3. Measurable disease according to RECIST v1.1 for all patients except patients with RET altered tumors; patients with RET altered tumors must have evaluable disease, but are not required to have measurable disease
4. Patients with treated, stable CNS metastases, including leptomeningeal carcinomatosis are allowed. The use of seizure prophylaxis is allowed. Patients requiring steroids must be at a stable or decreasing dose for at least 2 weeks prior to the start of RXDX-105 treatment.
5. Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2
6. Able to ingest oral medication
7. Other inclusion criteria apply

Exclusion Criteria for Phase 1b:

1. Treated with systemic anticancer therapy or an investigational agent within 2 weeks or 5 half-lives, whichever is shorter, prior to start of study drug treatment (4 weeks for antibody therapy and immunotherapy, and 2 weeks for bevacizumab in colon cancer patients)
2. Major surgery 21 days or less prior to starting study drug or has not recovered from adverse effects of such therapy
3. Radiotherapy within 2 weeks prior to start of study drug treatment (palliative radiation or stereotactic radiosurgery within 7 days prior to start of study treatment). Patients must have recovered from all radiotherapy-related toxicities
4. History of non-pharmacologically induced prolonged QTc interval (e.g., repeated demonstration of a QTc interval > 500 milliseconds from ECGs performed at least 24 hours apart)
5. Major active infection requiring parenteral antibiotics
6. Severe or unstable medical condition, such as congestive heart failure (New York Heart Association [NYHA] Class III or IV), ischemic heart disease, uncontrolled hypertension, uncontrolled diabetes mellitus, psychiatric condition, as well as an uncontrolled cardiac arrhythmia requiring medication (≥ Grade 2, according to NCI CTCAE v4.03), myocardial infarction within 6 months prior to starting study treatment, or any other significant or unstable concurrent medical illness that in the opinion of the Investigator would preclude protocol therapy
7. History of other previous cancer that would interfere with the determination of safety or efficacy of RXDX-105 with respect to the qualifying solid tumor malignancy
8. Known infection with human immunodeficiency virus (HIV) and active hepatitis B or hepatitis C
9. Current participation in another clinical study of an investigational agent, vaccine, or device. Concomitant participation in observational studies is acceptable
10. Presence of a significant gastrointestinal disorder that, in the opinion of the Investigator or Sponsor, could interfere with absorption of RXDX-105 (e.g., malabsorption syndrome, gastrointestinal surgery)
11. Known hypersensitivity to any of the components of RXDX-105

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 143 (Actual)
Dates: Start 2013-06; Primary Completion 2018-12 (Actual); Study Completion 2019-02 (Actual)

PRIMARY OUTCOMES:
Phase 1: Dose Limiting Toxicities | Approximately 12 months
  From signing of the informed consent up to approximately 12 months
Phase 1: Occurrence of Adverse Events | Approximately 12 months
  From signing of the informed consent up to approximately 12 months
Phase 1b: Occurrence of Adverse Events | Approximately 12 months
  To further assess the safety profile and tolerability of RXDX-105 at the RP2D

SECONDARY OUTCOMES:
Phase 1: Maximum observed plasma drug concentration (Cmax) | Day 1 to Day 16
Phase 1: Time of maximum observed plasma drug concentration (tmax) | Day 1 to Day 16
Phase 1: Area under the plasma drug concentration versus time curve from time 0 to infinity (AUC0-∞) | Day 1 to Day 16
Phase 1: Area under the plasma drug concentration versus time curve from time 0 to the last measureable drug concentration (AUC0-t) | Day 1 to Day 16
Phase 1: Area under the plasma drug concentration versus time curve from time 0 to 24 hours after study drug administration (AUC0-24) | Day 1 to Day 16
Phase 1: Terminal elimination rate constant (λz) | Day 1 to Day 16
Phase 1: Terminal elimination half-life (t1/2) | Day 1 to Day 16
Phase 1: Apparent clearance of study drug from plasma (CL/F) | Day 1 to Day 16
Phase 1b: Objective Response Rate | Approximately 12 months
  Objective response rate is defined as the proportion of patients with advanced solid tumors achieving best overall response of complete response (CR), or partial response (PR), as assessed using RECIST v1.1
Phase 1b: Duration of Objective Response | Approximately 12 months
  The duration of objective response is defined as the time interval from the date of first documented response (CR or PR) to disease progression or death, whichever occurs first
Phase 1b: Clinical Benefit Rate | Approximately 12 months
  Clinical benefit rate is defined as the proportion of patients achieving a complete response (CR), partial response (PR) or stable disease (SD) for 6 months

CONTACTS AND LOCATIONS:
Locations (14):
- United States (14):
  - City of Hope, Duarte, California
  - University of California Irvine College of Medicine, Irvine, California
  - University of California San Diego Moores Cancer Center, San Diego, California
  - Lombardi Comprehensive Cancer Center, Georgetown, Washington D.C., District of Columbia
  - Florida Cancer Center, Sarasota, Florida
  - University Cancer & Blood Center, LLC, Athens, Georgia
  - Massachusetts General Hospital/Beth Israel Deaconess Med. Ctr./Dana Farber Cancer Institute, Boston, Massachusetts
  - Henry Ford Health System, Detroit, Michigan
  - Karmanos Cancer Center, Detroit, Michigan
  - Washington University, St Louis, Missouri
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - University of Texas MD Anderson Cancer Center, Houston, Texas
  - University of Washington, Seattle Cancer Care Alliance, Seattle, Washington

REFERENCES:
- [Derived] Pietrantonio F, Di Nicolantonio F, Schrock AB, Lee J, Morano F, Fuca G, Nikolinakos P, Drilon A, Hechtman JF, Christiansen J, Gowen K, Frampton GM, Gasparini P, Rossini D, Gigliotti C, Kim ST, Prisciandaro M, Hodgson J, Zaniboni A, Chiu VK, Milione M, Patel R, Miller V, Bardelli A, Novara L, Wang L, Pupa SM, Sozzi G, Ross J, Di Bartolomeo M, Bertotti A, Ali S, Trusolino L, Falcone A, de Braud F, Cremolini C. RET fusions in a small subset of advanced colorectal cancers at risk of being neglected. Ann Oncol. 2018 Jun 1;29(6):1394-1401. doi: 10.1093/annonc/mdy090. PMID 29538669